CLINICAL TRIAL: NCT02994329
Title: Community-based Distribution of Oral HIV Self-testing Kits-A Pilot Intervention and Rapid Impact Evaluation
Brief Title: Community-based Distribution of Oral HIV Self-testing Kits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zambart (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIV-SELF 3IE
Record Dates: First submitted 2016-11-30; First posted 2016-12-15 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: HIV Seropositivity
Keywords: HIV testing; Linkage to care
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral HIV self test (Active Comparator): In this arm, community health workers conducting door-to-door HIV testing will offer oral HIV self testing (OraQuick® HIV Self-Test (Orasure Technologies, Thailand)) as an alternative to standard of care finger-prick HIV testing for individuals who are present at the time of the visit. In addition they will provide demonstration to an adult who is present at the time of the visit and leave up to 2 oral HIV self test kits to allow testing with the partner
  Interventions: Device: OraQuick® HIV Self-Test (Orasure Technologies, Thailand)
- Standard of Care (No Intervention): In this arm community health workers will conduct door-to-door HIV testing using the current Zambian national HIV testing algorithm of finger-prick rapid HIV tests

INTERVENTIONS:
Device: OraQuick® HIV Self-Test (Orasure Technologies, Thailand) — All individuals aged 16 and above who are approached by community health workers conducting door-to door HIV testing will be offered the choice to use an oral HIV self test kit or to have standard of care finger-prick rapid HIV testing
  Arms: Oral HIV self test

SUMMARY:
This cluster randomised trial aims to evaluate the impact of a pilot HIVST intervention of oral HIV self-testing (HIVST) as an option for HIV testing, in addition to the offer of home-based rapid HIV testing, through community health workers (CHW) on knowledge of HIV status among the general adult and adolescent population.

The primary outcome of the trial is the proportion of individuals who know their HIV status, defined as a self-report of being HIV positive or accepting testing (standard or self testing) from the CHW.

Embedded within the impact evaluation is a process evaluation that will explore the fidelity of the implementation of the intervention and outputs of the intervention. Qualitative data on actual use, management and disposal of the HIVST kits, acceptability of HIVST and any impacts on relationships (including between couples and with CHW) associated with use of HIVST kits.

DETAILED DESCRIPTION:
Trial Purpose This cluster randomised trial will evaluate the impact of a pilot intervention of oral HIV self-testing (HIVST) as an option for HIV testing, in addition to the offer of home-based rapid HIV testing, by community health workers (CHWs ) on knowledge of HIV status among the general adult and adolescent population.

Aim The overall aim of this trial is to investigate whether the inclusion of HIVST as an option for HIV testing, in addition to the offer of HIV testing with a finger-prick blood sample, increases the uptake of an offer of home-based HIV-testing overall relative to an offer of HIV testing with a finger-prick blood sample alone.

Secondary Objectives

1. Investigate whether the inclusion of HIVST as an option for HIV testing in addition to the offer of HIV testing with a finger-prick blood sample through CHW increases the uptake of an offer of HIV-testing among specific sub-populations including men, adolescents and individuals who have not previously tested relative to an offer of HIV testing with a finger-prick blood sample alone.
2. Investigate whether the inclusion of HIVST as an option for HIV testing in addition to the offer of HIV testing with a finger-prick blood sample through CHW increases the proportion of individuals' diagnosed HIV positive relative to an offer of HIV testing with a finger-prick blood sample alone.
3. Measure linkage to HIV treatment and care, or prevention services when HIVST is included as an option for HIV testing in addition to the offer of HIV testing with a finger-prick blood sample through CHW and levels of couples-testing.

Trial Design This cluster randomised trial will randomise community health worker zones (66 in total) to either distribute oral HIVST kits in addition to the offer of finger-prick rapid HIV testing (33 zones) or to offer finger-prick rapid HIV testing alone (33 zones). The trial is nested within theHPTN071/PopART trial and the CHWs to be randomised all work in 4 of the intervention sites of this study.

Trial location Four communities in the Copperbelt and Central province of Zambia have been chosen to participate in this trial.

Trial Participants All adults and adolescents aged 16 years or older living in these communities are eligible for participation if they consent to participate in the household visit and are eligible for HIV testing (individuals aged 16 years or older who do not report knowing their HIV status). The CHW will use the electronic data capture devices to collect all information.

Process Evaluation Measures and Data Collection Process evaluation data will be collected using standardised data collection forms developed for this trial, including forms to collect data on how many CHW attended training on the demonstration of HIVST and the number of HIVST kits procured. Data will also be collected on: 1). the number of households visited and offered the option of HIVST or door-to-door rapid finger-prick HIV testing, and follow-up visits to individuals receiving an HIVST kit(s). the number of community engagement activities performed to inform the community of the availability of HIVST kits. Data on number of households visited will be collected through the existing EDC devices with data on community activities collected from routine monitoring data. Expected outputs, namely the number of HIVST kits distributed for use by individuals present or absent at the time of the household visit, will also be collected through the existing EDC devices. Data on outcomes of interest will be collected through the existing EDC devices, with linkage data extracted using forms developed for HPTN071 and qualitative data collection, including the acceptability of HIVST and their distribution through CHW.

Measured as part of the Process Evaluation

The following measures will be estimated through qualitative and quantitative data collection as part of the process evaluation:

Inputs:How many CHW were trained to deliver the intervention? How many HIVST kits were procured? How many meetings with CABs, community mobilisers and other stakeholds were held? And how many attendees were at these meetings? Activities: How many door-to-door visits were conducted? How many communication activities were held in the communities? Outputs: How many HIVST kits were distributed? Were communities aware of the HIVST intervention and where to obtain HIVST kits?Was HIVST acceptable? How was it perceived by community members?

Ethical Considerations The trial will be conducted in accordance with Good Clinical Practice guidelines, and all research staff will receive GCP training. The Ethics Committees to approve this study will be the Biomedical Ethics Committee of the University of Zambia and the ethics committee of the London School of Hygiene and Tropical Medicine.

In all communities, HIV testing will follow the Zambian national HIV testing guidelines, with HIV testing services offered only to individuals aged 16 years or older and informed consent for HTS obtained as per the Ministry of Health guidelines. Individuals will be informed of the HTS process and have the right to decline HTS or provide written or verbal consent to HTS . For individuals absent at the time of the household visit, an index HIV testing client will be asked whether they agree to accept an HIVST on behalf of the absent household member and to provide a demonstration on how to perform the test to this same individual. This individual will be asked to sign an agreement statement, stating that they will only give the self-test kit to their spouse/partner. The absent individual can decline/opt-out of using the HIVST and this will be made clear to the individual accepting the HIVST.

Individuals who participate in any in-depth qualitative studies will be asked to provide written informed research consent.

Potential Harms Despite the increased availability of HIV testing services, including the door-to-door offer of home-based HIV testing, testing for HIV remains a sensitive issue subject to stigma and discrimination. HIV self-testing provides individuals more confidentiality and the opportunity to avoid the stigma of being seen to access HIV testing services at a clinic. Nonetheless, self-testing may pose harms distinct from facility- or community-based HIV testing strategies, including concerns of coercion to test.

To date, studies of the distribution of HIV self-tests by volunteer-counsellors in Malawi have found a low incidence of harms. Some 3% of individuals reported feeling coerced into self-testing, however, among this group of individuals, 92% were highly satisfied with self-testing and 94% stated they would recommend self-testing to family/friends.

Despite little evidence for social harms in other settings, offering a female an HIV self-test for her absent male partner may pose risks, including risk of gender based violence or coercion to self-test. The CHiPs are trained in providing couples HIV testing and counselling services and will only leave a self-test kit if it is clear that there is no history of violence in the relationship. Women will also be informed that the CHiP can return to counsel the couple on their HIV test result or to support conducting the oral HIV self-test. The CHiPs will also be trained to ensure that the person they leave the test kit with has demonstrated that they can read and understand the test instructions and are able to instruct others to properly conduct an HIV self-test. Further, the CHiPs will also ensure that the person they leave the test kit with understands the consequences of forced testing and acknowledges that they will not force anyone to test using the kit. To avoid inadvertent coercion by leaving an HIV self-test for an individual who refuses the offer of HIV-testing, a self-test will only be left for individuals who consent to have a self-test left for them.

ELIGIBILITY:
Inclusion Criteria:

* Resident in CHW zone
* Aged 16 years and above

Exclusion Criteria:

* age <16
* unable to provide informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8080 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
The proportion of the total resident adult population who know their HIV status | 3 Months
  Knowledge of know HIV status includes those individuals who self report to be HIV positive or who test using standard of care HIV tests or oral HIV self test kits with results reported

SECONDARY OUTCOMES:
Proportion of total resident adult population who consent to participate in the intervention | 3 Months
Proportion of male resident adult population who consent to participate in the intervention | 3 Months
  Outcome 2 restricted to men
Proportion of resident adult population who have previously not been reached by the PopART intervention who consent to participate in the intervention | 3 Months
  Outcome 2 restricted to those community members who have not previously been reached
Proportion of resident adolescent population who consent to participate in the intervention | 3 Months
  Outcome 2 restricted to adolescents aged 16-18 years
Proportion of all adults who consent to participate in the intervention who know their HIV status | 3 Months
  Knowledge of HIV status defined as perproportions of couples who primary outcome
Proportion of adults who test for HIV amongst those eligible for testing | 3 Months
  Eligibility for testing includes consent to participate in the intervention and not self-reporting being HIV positive
Proportion of couples who test for HIV and receive results as a couple | 3 Months
Factors associated with uptake of and experience with HIV self testing | 3 Months
  Qualitative data
Linkage to HIV prevention and care | 3 Months
Incremental cost effectiveness of the addition of oral HIV self testing into a package of door-to- door HIV testing provided by CHW | 3 Months
Reported social harms associated with HIV testing | 3 Months
  Social harms will be defined as any adverse event occurring as a direct result of HIV testing including domestic violence, marital break up or suicide. Social harms will be solicited by directly asking participants to report any events and also by passive reporting by community members, advisory boards or other bodies

CONTACTS AND LOCATIONS:
Overall Officials: Alwyn Mwinga, PhD, Principal Investigator — Zambart
Locations (1):
- Zambart, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
the de-identified data will be made available via International Initiative for Evaluation's (3ie) public access data repository.

REFERENCES:
- [Background] Hensen B, Lewis JJ, Schaap A, Tembo M, Mutale W, Weiss HA, Hargreaves J, Ayles H. Factors associated with HIV-testing and acceptance of an offer of home-based testing by men in rural Zambia. AIDS Behav. 2015 Mar;19(3):492-504. doi: 10.1007/s10461-014-0866-0. PMID 25096893
- [Background] Musheke M, Bond V, Merten S. Couple experiences of provider-initiated couple HIV testing in an antenatal clinic in Lusaka, Zambia: lessons for policy and practice. BMC Health Serv Res. 2013 Mar 14;13:97. doi: 10.1186/1472-6963-13-97. PMID 23496926
- [Background] Doyle AM, Mavedzenge SN, Plummer ML, Ross DA. The sexual behaviour of adolescents in sub-Saharan Africa: patterns and trends from national surveys. Trop Med Int Health. 2012 Jul;17(7):796-807. doi: 10.1111/j.1365-3156.2012.03005.x. Epub 2012 May 18. PMID 22594660
- [Derived] Mulubwa C, Hensen B, Phiri MM, Shanaube K, Schaap AJ, Floyd S, Phiri CR, Bwalya C, Bond V, Simwinga M, Mwenge L, Fidler S, Hayes R, Mwinga A, Ayles H; HPTN 071 (PopART) Study Team. Community based distribution of oral HIV self-testing kits in Zambia: a cluster-randomised trial nested in four HPTN 071 (PopART) intervention communities. Lancet HIV. 2019 Feb;6(2):e81-e92. doi: 10.1016/S2352-3018(18)30258-3. Epub 2018 Dec 21. PMID 30584047